CLINICAL TRIAL: NCT01307462
Title: Fluticasone Propionate, Azithromycin, and Montelukast Sodium in Treating Patients With Bronchiolitis Obliterans Who Previously Underwent Stem Cell Transplant
Brief Title: Targeted Therapy of Bronchiolitis Obliterans Syndrome
Acronym: FAM for BOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie Lee (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Stephanie Lee, Principal Investigator, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2367.00; NCI-2011-00203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA163438 (NIH); RDCRN 6503 (Other: DMCC)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Fluticasone; montelukast; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (BOS therapy) (Experimental): Patients receive fluticasone propionate inhaled PO BID, azithromycin PO 3 days a week, and montelukast sodium PO QD. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluticasone propionate; Drug: montelukast sodium; Drug: azithromycin

INTERVENTIONS:
Drug: fluticasone propionate — Given inhaled PO
  Other Names: Flonase; Flovent
Drug: montelukast sodium — Given PO
  Other Names: Singulair
Drug: azithromycin — Given PO
  Other Names: AzaSite; CP 62993; XZ-450

SUMMARY:
This phase II trial studies how well giving fluticasone propionate, azithromycin, and montelukast sodium (FAM) together works in treating patients with bronchiolitis obliterans who previously underwent stem cell transplant. FAM may be an effective treatment for bronchiolitis obliterans

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the combination treatment of FAM administered in post hematopoietic cell transplantation (HCT) recipients after the diagnosis of new onset bronchiolitis obliterans syndrome (BOS) can decrease the rate of treatment failure relative to an estimated historical rate of 40% using current therapies.

SECONDARY OBJECTIVES:

I. To confirm the safety profile of FAM.

II. To describe the effect on other standard pulmonary function test parameters: forced expiratory flow at 25%-75% of forced vital capacity (FVC) (FEF25-75), residual volume (RV), diffusion capacity of carbon monoxide (DLCO), forced expiratory volume in 1 second (FEV1)/FVC ratio and FEV1/slow vital capacity (SVC) ratio with FAM treatment.

III. To determine the change in molecular markers of inflammation and fibrosis in the blood with FAM treatment.

IV. To assess the impact of FAM on other chronic graft-versus-host disease (GVHD) manifestations.

V. To assess the impact of FAM on functional status, and health-related quality of life (HRQOL).

VI. To describe changes in steroid dosing.

OUTLINE:

Patients receive fluticasone propionate inhaled orally (PO) twice daily (BID), azithromycin PO 3 days a week, and montelukast sodium PO once daily (QD). Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BOS after HCT within the 6 months before study enrollment; for this study, BOS is defined as:

  * Forced expiratory volume in 1 second (FEV1) < 75% of the predicted normal and FEV1 to slow or inspiratory vital capacity ratio (FEV1/SVC or FEV1/IVC) =< 0.7, both measured before and after administration of bronchodilator OR
  * Pathologic diagnosis of BOS demonstrated by lung biopsy
* The baseline absolute FEV1 must be >= 10% lower than the pre-transplant absolute FEV1 as defined by the pre-transplant FEV1 minus the baseline FEV1, both measured before administration of a bronchodilator
* Participant (or parent/guardian) has the ability to understand and willingness to sign a written consent document

Exclusion Criteria:

* Recurrent or progressive malignancy requiring anticancer treatment
* Known history of allergy to or intolerance of montelukast, zafirlukast, azithromycin, erythromycin, or clarithromycin
* Pregnancy or nursing; all females of childbearing potential must have a negative serum or urine pregnancy test < 7 days before study drug administration
* Transaminases > 5 X upper limit of normal (ULN)
* Total bilirubin > 3 X ULN
* Chronic treatment with any inhaled steroid for > 1 month in the past three months
* Treatment with montelukast or zafirlukast for > 1 month during the past three months
* Treatment with prednisone at > 1.2 mg/kg/day (or equivalent steroid)
* Treatment with rifampin or phenobarbital, aspirin at doses > 325 mg/day, or ibuprofen at doses > 1200 mg/day
* Treatment with any Food and Drug Administration (FDA) non approved study medication within the past 4 weeks; off-label treatment with an FDA-approved medication is allowed
* Chronic oxygen therapy
* Evidence of any viral, bacterial or fungal infection involving the lung and not responding to appropriate treatment
* Clinical asthma (variable and recurring symptoms of airflow obstruction and bronchial hyper-responsiveness)
* Any condition that, in the opinion of the enrolling investigator, would interfere with the subject's ability to comply with the study requirements
* Uncontrolled substance abuse or psychiatric disorder
* Inability to perform pulmonary function tests (PFT) reliably, as determined by the enrolling investigator or PFT lab
* Life expectancy < 6 months at the time of enrollment as judged by the enrolling investigator
* Baseline post-bronchodilator FEV1 < 20% of predicted normal before or after albuterol

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium; Kirsten Williams, Study Chair — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - National Cancer Institute Experimental Transplantation & Immunology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
De-identified data are reported in aggregate.

REFERENCES:
- [Result] Williams KM, Cheng GS, Pusic I, Jagasia M, Burns L, Ho VT, Pidala J, Palmer J, Johnston L, Mayer S, Chien JW, Jacobsohn DA, Pavletic SZ, Martin PJ, Storer BE, Inamoto Y, Chai X, Flowers MED, Lee SJ. Fluticasone, Azithromycin, and Montelukast Treatment for New-Onset Bronchiolitis Obliterans Syndrome after Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2016 Apr;22(4):710-716. doi: 10.1016/j.bbmt.2015.10.009. Epub 2015 Oct 22. PMID 26475726
- [Derived] Inamoto Y, Martin PJ, Onstad LE, Cheng GS, Williams KM, Pusic I, Ho VT, Arora M, Pidala J, Flowers MED, Gooley TA, Lawler RL, Hansen JA, Lee SJ. Relevance of Plasma Matrix Metalloproteinase-9 for Bronchiolitis Obliterans Syndrome after Allogeneic Hematopoietic Cell Transplantation. Transplant Cell Ther. 2021 Sep;27(9):759.e1-759.e8. doi: 10.1016/j.jtct.2021.06.006. Epub 2021 Jun 12. PMID 34126278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (BOS Therapy)
Started | 36
Completed | 35
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 57 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Failed Treatment
Description: Treatment failure is defined as sustained, absolute decrease (worsening) of the FEV1 by >= 10% predicted in comparison to the baseline FEV1. Must be confirmed by a second PFT 2 weeks after the first measurement.
Time Frame: Within 3 months after initiation of study medications
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 36
Participants | 2

2. Secondary Outcome: Number of Subjects Who Experienced Grade 3-5 SAEs Attributable to FAM and Number of Subjects Who Stopped FAM as a Result
Description: National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) (v4.0)
Time Frame: From baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 36
Participants
  SAEs attributable to FAM | 11
  Stopped FAM during study | 1

3. Secondary Outcome: Number of Subjects Who Experienced Statistically Significant Changes in FVC, TLC, RV, DLCO
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 36
Participants | 0

4. Secondary Outcome: Changes in Blood Molecular Markers: IL8 (Azithromycin), Cysteinyl and LTB4 (Monteleukast), and IL1B, TNF, and IL6, as Well as Neutrophil Count (Fluticasone)
Time Frame: Baseline to 6 months
Population: Data were not collected
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Subjects With Improvements in Other Chronic GVHD Characteristics
Description: Only includes subjects who had complete or partial response according to the National Institute of Health (NIH) consensus criteria.
Time Frame: Baseline and 3 months
Population: 33 of 36 participants were evaluable at 3 months due to missing provider survey data
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 33
Participants | 12

6. Secondary Outcome: Number of Subjects Were Able to Reduce Their Systemic Steroid Exposure by >=50%
Time Frame: Baseline to 6 months
Population: 24 out of 36 subjects were evaluable at 6mo due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 24
Participants | 17

7. Secondary Outcome: Changes in Symptoms as Measured by Patient Self-report--Short Form-36 (SF-36)
Description: SF-36 subscales have min=0 and max=100; results are given as change in 6mo score compared to baseline score, not actual score, and a positive change is correlated with improvement in clinical outcome.
Time Frame: Baseline and 6 months
Population: 24 of 36 subjects were evaluable at 6mo due to missing patient survey data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 24
units on a scale
  SF-36 norm-based physical functioning score | 0.0 [-23.15 to 14.73]
  SF-36 norm-based role-physical score | 0.0 [-17.14 to 39.18]
  SF-36 norm-based bodily pain score | 0.0 [-13.52 to 17.33]
  SF-36 norm-based general health score | -2.38 [-20.02 to 17.64]
  SF-36 norm-based vitality score | 1.56 [-15.61 to 21.85]
  SF-36 norm-based social functioning score | 5.45 [-27.27 to 38.18]
  SF-36 norm-based role-emotional score | 0.0 [-23.32 to 23.32]
  SF-36 norm-based mental health score | 0.0 [-11.26 to 16.9]
  SF-36 standardized physical component score | -1.21 [-21.65 to 25.16]
  SF-36 standardized mental component score | 1.64 [-21.63 to 25.76]
Statistical Analysis 1: Comparison: Treatment (BOS Therapy); SF-36 norm-based physical functioning score; Test type: Superiority; p = .81, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Treatment (BOS Therapy); SF-36 norm-based role-physical score; Test type: Superiority; p = .18, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Treatment (BOS Therapy); SF-36 norm-based bodily pain score; Test type: Superiority; p = .48, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Treatment (BOS Therapy); SF-36 norm-based general health score; Test type: Superiority; p = .26, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Treatment (BOS Therapy); SF-36 norm-based vitality score; Test type: Superiority; p = .23, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Treatment (BOS Therapy); SF-36 norm-based social functioning score; Test type: Superiority; p = .36, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Treatment (BOS Therapy); SF-36 norm-based role-emotional score; Test type: Superiority; p = .41, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Treatment (BOS Therapy); SF-36 norm-based mental health score; Test type: Superiority; p = .80, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Treatment (BOS Therapy); SF-36 standardized physical component score; Test type: Superiority; p = .80, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Treatment (BOS Therapy); SF-36 standardized mental component score; Test type: Superiority; p = .23, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Changes in Symptoms as Measured by Patient Self-report--Functional Assessment of Chronic Illness Therapy (FACT)
Description: FACT-BMT subscales have various min/max, see below; results are given as change in 6mo score compared to baseline score, not actual score, and a positive change is correlated with improvement in clinical outcome.
  FACT physical well-being (0-28) FACT social/family well-being (0-28) FACT emotional well-being (0-24) FACT functional well-being (0-28) FACT Bone Marrow Transplant (BMT) subscale (0-40) FACT trial outcome index (0-96) FACT-General (G) (0-108) FACT-BMT total (0-148)
Time Frame: Baseline and 6 months
Population: 24 of 36 subjects were evaluable at 6mo due to missing patient survey data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 24
units on a scale
  FACT physical well-being | 0.5 [-8 to 12]
  FACT social/family well-being | -1 [-6.83 to 7]
  FACT emotional well-being | 0 [-6 to 17]
  FACT functional well-being | 1 [-15 to 13]
  FACT BMT subscale | -0.78 [-7 to 10]
  FACT trial outcome index | 2 [-30 to 22]
  FACT-G | 2.5 [-23 to 23.67]
  FACT-BMT total | 2.17 [-30 to 25]
Statistical Analysis 1: Comparison: Treatment (BOS Therapy); FACT physical well-being; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Treatment (BOS Therapy); FACT social/family well-being; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Treatment (BOS Therapy); FACT emotional well-being; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Treatment (BOS Therapy); FACT functional well-being; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Treatment (BOS Therapy); FACT BMT subscale; Test type: Superiority; p = .84, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Treatment (BOS Therapy); FACT trial outcome index; Test type: Superiority; p = .37, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Treatment (BOS Therapy); FACT-G; Test type: Superiority; p = .71, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Treatment (BOS Therapy); FACT-BMT total; Test type: Superiority; p = .54, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Changes in Symptoms as Measured by Patient Self-report--Human Activities Profile (HAP)
Description: HAP subscales have min=0 and max=94; results are given as change in 6mo score compared to baseline score, not actual score, and a positive change is correlated with improvement in clinical outcome.
  Maximum Activity Score (MAS) is highest item number answered still doing. Represents highest oxygen demanding activity that respondent still performs.
  Adjusted Activity Score (AAS) is MAS minus total number of stopped doing responses below MAS. A measure of usual daily activities.
  Modified AAS is MAS minus total number of stopped doing responses below MAS but not penalized for not doing activities not permitted post transplant. The following items are not counted against the score:11,15,19,20,22,25,34,41,42,47,49,50,52,53,54,57,72,73,77,78.
Time Frame: Baseline and 6 months
Population: 24 of 36 subjects were evaluable at 6mo due to missing patient survey data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 24
units on a scale
  HAP MAS | 0.5 [-41 to 30]
  HAP AAS | 4.5 [-49 to 42]
  Modified HAP AAS | 3.5 [-46 to 36]
Statistical Analysis 1: Comparison: Treatment (BOS Therapy); HAP maximum activity score - highest item still doing; Test type: Superiority; p = .37, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Treatment (BOS Therapy); HAP adjusted activity score - MAS minus stopped; Test type: Superiority; p = .39, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Treatment (BOS Therapy); Modified HAP adjusted activity score; Test type: Superiority; p = .39, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Changes in Symptoms as Measured by Patient Self-report--Lee Chronic GVHD Symptom Scale
Description: Lee symptom scale (LSS) has subscales with min=0, max=100; results are given as change in 6mo score compared to baseline score, not actual score, and a negative change is correlated with improvement in clinical outcome.
Time Frame: Baseline and 6 months
Population: 24 of 36 subjects were evaluable at 6mo due to missing patient survey data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (BOS Therapy)
Number analyzed (Participants) | 24
units on a scale
  LSS skin scale | -5.63 [-45 to 50]
  LSS energy scale | -7.14 [-39.29 to 14.29]
  LSS lung scale | -5 [-55 to 45]
  LSS eye scale | -8.33 [-66.67 to 8.33]
  LSS nutrition scale | 0 [-30 to 10]
  LSS psychological scale | 0 [-50 to 50]
  LSS mouth scale | 0 [-75 to 0]
  LSS overall summary scale | -7.77 [-32.21 to 2.52]
Statistical Analysis 1: Comparison: Treatment (BOS Therapy); Lee symptom skin scale; Test type: Superiority; p = .11, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Treatment (BOS Therapy); Lee symptom energy scale; Test type: Superiority; p = .007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Treatment (BOS Therapy); Lee symptom lung scale; Test type: Superiority; p = .20, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Treatment (BOS Therapy); Lee symptom eye scale; Test type: Superiority; p = .002, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Treatment (BOS Therapy); Lee symptom nutrition scale; Test type: Superiority; p = .52, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Treatment (BOS Therapy); Lee symptom psychological scale; Test type: Superiority; p = .22, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Treatment (BOS Therapy); Lee symptom mouth scale; Test type: Superiority; p = .002, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Treatment (BOS Therapy); Lee symptom overall summary scale; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment (BOS Therapy)
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 24/36
Other Adverse Events (participants affected / at risk) | 9/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (BOS Therapy) (N=36)
Edema limbs (General disorders) | 1 (1)
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fluid overload (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (BOS Therapy) (N=36)
Cavitary Pulmonary Lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No